CLINICAL TRIAL: NCT00615056
Title: A Randomized, Phase 2 Study Of FOLFOX Or FOLFIRI With AG-013736 Or Bevacizumab (Avastin) In Patients With Metastatic Colorectal Cancer After Failure Of An Irinotecan Or Oxaliplatin-Containing First-Line Regimen
Brief Title: A Study Combining FOLFOX or FOLFIRI With AG-013736 or Bevacizumab (Avastin) in Patients With Metastatic Colorectal Cancer After Failure Of One First Line Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4061034
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Results first posted 2012-04-20 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Irinotecan; Leucovorin; Fluorouracil; Axitinib; Folfox protocol; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- B (Active Comparator): Bevacizumab (avastin)
  Interventions: Drug: Bevacizumab (avastin); Drug: FOLFIRI (Irinotecan, leucovorin, 5-fluorouracil [5FU])
- C (Experimental): AG-013736 (axitinib)
  Interventions: Drug: AG-013736 (axitinib); Drug: FOLFOX (oxaliplatin, leucovorin, 5-fluorouracil [5FU])
- A (Experimental): AG-013736 (axitinib)
  Interventions: Drug: AG-013736 (axitinib); Drug: FOLFIRI (irinotecan, leucovorin, 5-fluorouracil [5FU])
- D (Active Comparator): bevacizumab (avastin)
  Interventions: Drug: Bevacizumab (avastin); Drug: FOLFOX (oxaliplatin, leucovorin, 5-fluorouracil [5FU])

INTERVENTIONS:
Drug: Bevacizumab (avastin) — Bevacizumab intravenous [IV] infusion 5 mg/kg every two weeks until disease progression, intolerance or withdrawal of consent.
  Arms: B
Drug: FOLFIRI (Irinotecan, leucovorin, 5-fluorouracil [5FU]) — Irinotecan (180 mg/m²) intravenous infusion [IV] over 90 minutes, concurrently with leucovorin (400 mg/m²) intravenous infusion [IV] over 2 hours followed immediately by 5-FU bolus (400 mg/m²) intravenous [IV] and a subsequent 5-FU infusion (2400 mg/m² over 46-48 hours), repeated every 2 weeks until disease progression, intolerance or withdrawal of consent.
  Arms: B
Drug: AG-013736 (axitinib) — Axitinib is given at a starting dose of 5 mg twice daily [BID] continuous dosing until disease progression, intolerance or withdrawal of consent.
  Arms: C
Drug: FOLFOX (oxaliplatin, leucovorin, 5-fluorouracil [5FU]) — Oxaliplatin (85 mg/m²) intravenous infusion [IV] over 120 minutes, concurrently with leucovorin (400 mg/m²) intravenous infusion [IV] over 2 hours followed by 5-FU IV bolus (400 mg/m²) and a subsequent 5-FU IV infusion (2400 mg/m² over 46-48 hours), repeated every 2 weeks until disease progression, intolerance or withdrawal of consent.
  Arms: C
Drug: AG-013736 (axitinib) — Axitinib is given at a starting dose of 5 mg twice daily [BID] continuous dosing until disease progression, intolerance or withdrawal of consent.
  Arms: A
Drug: FOLFIRI (irinotecan, leucovorin, 5-fluorouracil [5FU]) — Irinotecan (180 mg/m²) intravenous infusion [IV] over 90 minutes, concurrently with leucovorin (400 mg/m²) intravenous infusion [IV] over 2 hours followed immediately by 5-FU bolus (400 mg/m²) IV and a subsequent 5-FU IV infusion (2400 mg/m² over 46-48 hours), repeated every 2 weeks until disease progression, intolerance or withdrawal of consent.
  Arms: A
Drug: Bevacizumab (avastin) — Bevacizumab intravenous infusion [IV] 5 mg/kg every two weeks until disease progression, intolerance or withdrawal of consent.
  Arms: D
Drug: FOLFOX (oxaliplatin, leucovorin, 5-fluorouracil [5FU]) — Oxaliplatin (85 mg/m²) IV infusion over 120 minutes, concurrently with leucovorin (400 mg/m²) intravenous infusion [IV] over 2 hours followed by 5-FU IV bolus (400 mg/m²) and a subsequent 5-FU IV infusion (2400 mg/m² over 46-48 hours), repeated every 2 weeks until disease progression, intolerance or withdrawal of consent.
  Arms: D

SUMMARY:
The study is designed to demonstrate that the combination of AG-013736 with either FOLFIRI or FOLFOX is superior to FOLFIRI or FOLFOX in combination with bevacizumab (Avastin) in delaying tumor progression in the second-line treatment of patients with metastatic colorectal cancer after failure of an irinotecan or oxaliplatin-containing first-line regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented colorectal cancer plus one of the following:
* Failure of one prior irinotecan- or oxaliplatin-containing regimen, or
* Adjuvant refractory to irinotecan- or oxaliplatin-containing regimen.

Exclusion Criteria:

* Prior treatment in first line metastatic setting with more than one regimen
* Prior irradiation of more than 25% of bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- United States (42):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Antioch, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Pleasant Hill, California
  - Pfizer Investigational Site, San Leandro, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Bonita Springs, Florida
  - Pfizer Investigational Site, Bradenton, Florida
  - Pfizer Investigational Site, Cape Coral, Florida
  - Pfizer Investigational Site, Englewood, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Port Charlotte, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Venice, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Ringgold, Georgia
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Paducah, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, New Albany, Mississippi
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Fairfield, Ohio
  - Pfizer Investigational Site, Hamilton, Ohio
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Hixson, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Paris, Tennessee
  - Pfizer Investigational Site, Smyrna, Tennessee
  - Pfizer Investigational Site, Union City, Tennessee
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Mechanicsville, Virginia
  - Pfizer Investigational Site, Midlothian, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
- Canada (3):
  - Pfizer Investigational Site, Greenfield Park, Quebec
  - Pfizer Investigational Site, Lévis, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- France (4):
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Villejuif
- Italy (3):
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Roma
- Japan (3):
  - Pfizer Investigational Site, Kashiwa, Chiba
  - Pfizer Investigational Site, Suntougun, Shizuoka
  - Pfizer Investigational Site, Chuo-ku, Tokyo
- Pfizer Investigational Site, Warsaw, Poland
- South Korea (3):
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Jeollanam-do
  - Pfizer Investigational Site, Seoul
- Spain (3):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061034&StudyName=A%20Study%20Combining%20FOLFOX%20or%20FOLFIRI%20with%20AG-013736%20or%20Bevacizumab%20%28Avastin%29%20in%20Patients%20with%20Metastatic%20Colorectal%20Cancer%20After%20Failur

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib + FOLFIRI: Axitinib (AG-013736) tablet starting dose 5 milligram (mg) orally twice daily (BID) along with combination chemotherapy of irinotecan, 5- flurouracil (5-FU) and leucovorin (LV) (FOLFIRI) regimen consisting of irinotecan 180 mg per square meter (mg/m^2) 90 minutes intravenous (IV) infusion, concurrently with LV 400 mg/m^2 (or levo-leucovarin [l-LV] 200 mg /m^2) 2 hours (hrs) IV infusion followed immediately by 5-FU 400 mg/m^2 IV bolus injection and a subsequent 5-FU 2400 mg/m^2 46-48 hrs IV infusion on Day 1 of each 2 week cycle.
- Bevacizumab + FOLFIRI: Bevacizumab 5mg/kilogram (kg) 30-90 minutes IV infusion (based on tolerance) every 2 weeks along with FOLFIRI regimen consisting of irinotecan 180 mg/m^2 90 minutes IV infusion, concurrently with LV 400 mg/m^2 (or l-LV 200 mg /m^2) 2 hrs IV infusion followed immediately by 5-FU 400 mg/m^2 IV bolus injection and a subsequent 5-FU 2400 mg/m^2 46-48 hrs IV infusion on Day 1 of each 2 week cycle.
- Axitinib + FOLFOX: Axitinib (AG-013736) tablet starting dose 5 mg BID along with combination chemotherapy of oxaliplatin, LV and 5-FU (FOLFOX) regimen consisting of oxaliplatin 85 mg/m^2 120 minutes IV infusion, concurrently with LV 400 mg/m^2 (or l-LV 200 mg /m^2) 2 hrs IV infusion followed immediately by 5-FU 400 mg/m^2 IV bolus injection and a subsequent 5-FU 2400 mg/m^2 46-48 hrs IV infusion on Day 1 of each 2 week cycle.
- Bevacizumab + FOLFOX: Bevacizumab 5mg/kg 30-90 minutes IV infusion (based on tolerance) every 2 weeks along with FOLFOX regimen consisting of oxaliplatin 85 mg/m^2 120 minutes IV infusion, concurrently with LV 400 mg/m^2 (or l-LV 200 mg /m^2) 2 hrs IV infusion followed immediately by 5-FU 400 mg/m^2 IV bolus injection and a subsequent 5-FU 2400 mg/m^2 46-48 hrs IV infusion on Day 1 of each 2 week cycle.
Period: Overall Study
Arm/Group | Axitinib + FOLFIRI | Bevacizumab + FOLFIRI | Axitinib + FOLFOX | Bevacizumab + FOLFOX
Started | 49 | 51 | 36 | 35
Treated | 46 | 51 | 36 | 35
Completed | 0 | 0 | 0 | 0
Not Completed | 49 | 51 | 36 | 35
Not completed — Death | 31 | 31 | 21 | 23
Not completed — Lost to Follow-up | 1 | 2 | 4 | 5
Not completed — Other | 13 | 15 | 10 | 7
Not completed — Objective progression or relapse | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Discontinued by Sponsor | 1 | 0 | 0 | 0
Not completed — Randomized but not treated | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Axitinib + FOLFIRI | Bevacizumab + FOLFIRI | Axitinib + FOLFOX | Bevacizumab + FOLFOX | Total
Number analyzed (Participants) | 49 | 51 | 36 | 35 | 171
Age, Customized [Number; unit: Participants]
  18 to 44 years | 5 | 6 | 3 | 1 | 15
  45 to 64 years | 30 | 34 | 21 | 22 | 107
  Greater than and equal to 65 years | 14 | 11 | 12 | 12 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 24 | 20 | 11 | 73
  Male | 31 | 27 | 16 | 24 | 98

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time in months from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.4. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline until disease progression or discontinuation from the study due to any cause, assessed every 8 week up to 130 weeks
Population: Intent-to-treat (ITT) population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug, or receive a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + FOLFIRI | Bevacizumab + FOLFIRI | Axitinib + FOLFOX | Bevacizumab + FOLFOX
Number analyzed (Participants) | 49 | 51 | 36 | 35
Months | 5.72 [4.50 to 7.42] | 6.87 [4.96 to 9.13] | 7.59 [5.62 to 11.07] | 6.44 [5.52 to 13.11]
Statistical Analysis 1: Comparison: Axitinib + FOLFIRI vs Bevacizumab + FOLFIRI; Differences in PFS between treatment arms was analyzed by 1-sided log rank test, stratified for Eastern Cooperative Oncology Group (ECOG) performance status (0 versus 1) and prior treatment with bevacizumab (yes versus no); Test type: Superiority or Other; p = 0.8268, Log Rank — One-sided log-rank test at alpha = 0.15 significance level was used; Hazard Ratio (HR) = 1.273, 95% CI 2-sided [0.769 to 2.108]
Statistical Analysis 2: Comparison: Axitinib + FOLFOX vs Bevacizumab + FOLFOX; Differences in PFS between treatment arms was analyzed by 1-sided log rank test, stratified for ECOG performance status (0 versus 1) and prior treatment with bevacizumab (yes versus no); Test type: Superiority or Other; p = 0.5498, Log Rank — One-sided log-rank test at alpha = 0.15 significance level was used; Hazard Ratio (HR) = 1.041, 95% CI 2-sided [0.553 to 1.041]

2. Secondary Outcome: Overall Survival (OS)
Description: Time in months from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 30.4. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline until death or up to 1 year after the randomization of last participant
Population: ITT population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug, or receive a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + FOLFIRI | Bevacizumab + FOLFIRI | Axitinib + FOLFOX | Bevacizumab + FOLFOX
Number analyzed (Participants) | 49 | 51 | 36 | 35
Months | 12.9 [10.2 to 16.6] | 15.7 [12.1 to 23.0] | 17.1 [10.1 to 23.0] | 14.1 [9.0 to 16.4]
Statistical Analysis 1: Comparison: Axitinib + FOLFIRI vs Bevacizumab + FOLFIRI; Differences in OS between treatment arms was analyzed by 1-sided log rank test, stratified for ECOG performance status (0 versus 1) and prior treatment with bevacizumab (yes versus no); Test type: Superiority or Other; p = 0.8828, Log Rank — One-sided log-rank test at alpha = 0.15 significance level was used; Hazard Ratio (HR) = 1.355, 95% CI 2-sided [0.820 to 2.238]
Statistical Analysis 2: Comparison: Axitinib + FOLFOX vs Bevacizumab + FOLFOX; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1159, Log Rank — One-sided log-rank test at alpha = 0.15 significance level was used; Hazard Ratio (HR) = 0.689, 95% CI 2-sided [0.373 to 1.273]

3. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. PR are those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent.
Time Frame: Baseline until disease progression or discontinuation from the study due to any cause, assessed every 8 weeks up to 130 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib + FOLFIRI | Bevacizumab + FOLFIRI | Axitinib + FOLFOX | Bevacizumab + FOLFOX
Number analyzed (Participants) | 49 | 51 | 36 | 35
Percentage of participants | 24.5 [13.3 to 38.9] | 23.5 [12.8 to 37.5] | 19.4 [8.2 to 36.0] | 20.0 [8.4 to 36.9]
Statistical Analysis 1: Comparison: Axitinib + FOLFIRI vs Bevacizumab + FOLFIRI; One-sided Pearson chi square test at alpha = 0.15 significance level was used; Test type: Superiority or Other; p = 0.4552, Chi-squared; Mean Difference (Final Values) = 1, 95% CI 2-sided [-15.8 to 17.7]
Statistical Analysis 2: Comparison: Axitinib + FOLFOX vs Bevacizumab + FOLFOX; One-sided Pearson chi square test at alpha = 0.15 significance level was used; Test type: Superiority or Other; p = 0.5235, Chi-squared; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-19.1 to 18.0]

4. Secondary Outcome: Duration of Response (DR)
Description: Time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.4. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 3
Population: DR was calculated for the subgroup of participants from the ITT set, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + FOLFIRI | Bevacizumab + FOLFIRI | Axitinib + FOLFOX | Bevacizumab + FOLFOX
Number analyzed (Participants) | 12 | 12 | 7 | 7
Months | 7.52 [5.22 to NA] — Upper limit of confidence interval was not estimable due to the large number of participants censored. | 12.29 [7.39 to 12.84] | 10.15 [4.17 to 12.91] | 10.94 [4.53 to 12.68]

5. Secondary Outcome: Change From Baseline in MD Anderson Symptoms Inventory Diarrhea (MDASI-D) Symptom Severity Score at Day 1 of Cycles 2-5, Day 1 of Every Odd-numbered Cycle Throughout the Study and End of Treatment (Cycle 65) or Withdrawal
Description: Symptom severity score is comprised of average of 14 MDASI-D core items (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, remembering things, lack of appetite, drowsiness, dry mouth, sadness, vomiting, numbness or tingling and diarrhea) and ranges from 0 to 10. Participants were asked to rate severity of each symptom at their worst in last week; each item rated from 0 to 10, with 0 = symptom not present and 10 = as bad as you can imagine. Lower scores indicated better outcome. Total average score range: 0 to 10.
Time Frame: Baseline, Day 1 of cycles 2- 5, Day 1 of every odd-numbered cycle throughout the study and end of treatment (cycle 65) or withdrawal
Population: ITT population. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' is number of participants analyzed at specific time point for each treatment arm respectively.
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Axitinib + FOLFIRI | Bevacizumab + FOLFIRI | Axitinib + FOLFOX | Bevacizumab + FOLFOX
Number analyzed (Participants) | 39 | 46 | 35 | 33
Units on a Scale
  Baseline (n=39,46,35,33) | 2.1 [1.6 to 2.6] | 1.8 [1.3 to 2.2] | 1.9 [1.3 to 2.5] | 2.0 [1.4 to 2.7]
  Change at Cycle 2/Day 1 (n=35, 39, 34,28) | 0.6 [0.2 to 1.1] | 0.5 [-0.1 to 1.0] | 0.7 [0.2 to 1.2] | 0.0 [-0.4 to 0.5]
  Change at Cycle 3/Day 1 (n=36,36,33,26) | 0.8 [0.2 to 1.4] | 0.2 [-0.3 to 0.6] | 0.3 [-0.4 to 1.0] | 0.2 [-0.3 to 0.7]
  Change at Cycle 4/Day 1 (n=29,37,32,25) | 0.8 [0.0 to 1.5] | 0.0 [-0.4 to 0.5] | 0.5 [-0.2 to 1.1] | 0.5 [-0.1 to 1.1]
  Change at Cycle 5/Day 1 (n=28,29,24,24) | 0.5 [0.0 to 1.1] | 0.1 [-0.4 to 0.7] | 0.9 [0.2 to 1.7] | 0.4 [-0.2 to 0.9]
  Change at Cycle 7/Day 1 (n=26,31,22,20) | 0.7 [0.1 to 1.2] | 0.0 [-0.6 to 0.5] | 0.6 [0.1 to 1.1] | 0.2 [-0.5 to 0.9]
  Change at Cycle 9/Day 1 (n=19,26,19,17) | 1.1 [0.3 to 1.9] | -0.2 [-0.7 to 0.2] | 0.6 [-0.1 to 1.3] | 0.8 [0.3 to 1.3]
  Change at Cycle 11/Day 1 (n=15,24,16,15) | 1.0 [0.1 to 1.9] | 0.1 [-0.5 to 0.7] | 1.0 [0.2 to 1.8] | 0.1 [-0.8 to 1.1]
  Change at Cycle 13/Day 1 (n=13,19,15,10) | 1.0 [-0.5 to 2.6] | 0.1 [-0.6 to 0.7] | 0.9 [0.2 to 1.6] | 0.8 [0.1 to 1.4]
  Change at Cycle 15/Day 1 (n=7,17,12,8) | 0.8 [-1.6 to 3.3] | 0.2 [-0.3 to 0.7] | 0.5 [-0.4 to 1.3] | 1.0 [0.4 to 1.6]
  Change at Cycle 17/Day 1 (n=6,11,11,7) | 2.0 [-0.9 to 5.0] | 0.4 [-0.3 to 1.0] | 0.9 [0.1 to 1.8] | 1.7 [0.7 to 2.7]
  Change at Cycle 19/Day 1 (n=6,10,9,5) | 1.3 [-1.5 to 4.1] | 0.5 [-0.7 to 1.7] | 0.8 [-0.2 to 1.8] | 1.4 [0.7 to 2.2]
  Change at Cycle 21/Day 1 (n=6,9,7,4) | 1.1 [-2.2 to 4.4] | 0.5 [-0.5 to 1.5] | 0.9 [-0.9 to 2.7] | 1.6 [0.3 to 2.8]
  Change at Cycle 23/Day 1 (n=5,7,6,4) | 2.6 [0.3 to 4.8] | -0.3 [-0.9 to 0.3] | 0.4 [-1.4 to 2.3] | 1.0 [0.8 to 1.2]
  Change at Cycle 25/Day 1 (n=5,7,6,3) | 2.2 [-1.2 to 5.6] | 0.1 [-1.2 to 1.4] | 0.2 [-2.0 to 2.3] | 1.0 [0.5 to 1.4]
  Change at Cycle 27/Day 1 (n=2,7,3,3) | 2.3 [-20.8 to 25.5] | 0.4 [-1.4 to 2.3] | 0.3 [-5.4 to 5.9] | 1.1 [0.6 to 1.5]
  Change at Cycle 29/Day 1 (n=2,5,2,3) | 2.8 [-25.8 to 31.4] | -0.2 [-1.3 to 0.9] | -0.8 [-1.7 to 0.1] | 0.9 [-0.3 to 2.1]
  Change at Cycle 31/Day 1 (n=1,5,2,2) | 4.9 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | -0.4 [-1.2 to 0.3] | -0.3 [-5.7 to 5.2] | 0.9 [-1.4 to 3.2]
  Change at Cycle 33/Day 1 (n=1,3,2,1) | 5.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | -0.6 [-3.2 to 2.0] | -0.8 [-7.6 to 6.1] | 0.5 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 35/Day 1 (n=0,4,1,1) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.4 [-1.5 to 0.7] | 0.4 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 2.4 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 37/Day 1 (n=0,4,0,1) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.5 [-1.3 to 0.4] | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 1.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 39/Day 1 (n=0,2,0,1) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.4 [-0.8 to 0.1] | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 1.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 41/Day 1 (n=0,2,0,1) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [-0.8 to 0.1] | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 1.4 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 43/Day 1 (n=0,1,0,1) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.4 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 2.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 45/Day 1 (n=0,0,0,1 ) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 2.2 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 47/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.4 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 49/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.5 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 51/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.4 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 53/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.4 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 55/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 57/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 59/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 61/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.2 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 63/Day 1 (n=0,0,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 65/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.4 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at end of treatment (n=21,29,27,22) | 0.7 [-0.2 to 1.6] | 0.5 [-0.1 to 1.0] | 1.3 [0.4 to 2.1] | 0.9 [0.1 to 1.7]

6. Secondary Outcome: Change From Baseline in MDASI-D Symptom Interference Score at Day 1 of Cycles 2-5, Day 1 of Every Odd-numbered Cycle Throughout the Study and End of Treatment (Cycle 65) or Withdrawal
Description: Symptom Interference score is comprised of the average of 6 items on feeling or function from the MDASI-D core (general activity, mood, work, relations with others, walking, and enjoyment of life) and ranges from 0 to 10. Participants were asked to rate how much symptoms have interfered in last week; each item rated from 0 to 10, with 0 = did not interfere and 10 = interfered completely. Lower scores indicated better outcome. Total average score range: 0 to 10.
Time Frame: Baseline, Day 1 of cycle 2-5, Day 1 of every odd-numbered cycle throughout the study and end of treatment (cycle 65) or withdrawal
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Axitinib + FOLFIRI | Bevacizumab + FOLFIRI | Axitinib + FOLFOX | Bevacizumab + FOLFOX
Number analyzed (Participants) | 39 | 46 | 35 | 33
Units on a Scale
  Baseline (n=39,46,35,33) | 2.1 [1.4 to 2.8] | 1.7 [1.1 to 2.3] | 2.4 [1.6 to 3.2] | 2.8 [1.8 to 3.9]
  Change at Cycle 2/Day 1 (n=35, 39, 34, 28) | 0.8 [0.0 to 1.5] | 0.9 [0.2 to 1.6] | 0.1 [-0.6 to 0.7] | -0.5 [-1.2 to 0.1]
  Change at Cycle 3/Day 1 (n=36,36,33,26) | 1.3 [0.5 to 2.2] | 0.3 [-0.3 to 0.8] | 0.3 [-0.6 to 1.2] | -0.2 [-1.0 to 0.6]
  Change at Cycle 4/Day 1 (n=29,37,32,25) | 0.8 [-0.1 to 1.7] | -0.2 [-0.9 to 0.4] | 0.2 [-0.6 to 1.1] | 0.5 [-0.2 to 1.3]
  Change at Cycle 5/Day 1 (n=28,29,24,24) | 1.0 [0.3 to 1.6] | 0.4 [-0.7 to 1.4] | 0.8 [-0.4 to 2.0] | 0.3 [-0.6 to 1.2]
  Change at Cycle 7/Day 1 (n=26,30,22,20) | 0.7 [-0.1 to 1.5] | 0.4 [-0.4 to 1.2] | 0.4 [-0.3 to 1.1] | 0.0 [-0.8 to 0.7]
  Change at Cycle 9/Day 1 (n=18,25,19,17) | 1.1 [0.2 to 1.9] | 0.3 [-0.6 to 1.1] | 0.6 [-0.5 to 1.6] | 0.3 [-0.8 to 1.4]
  Change at Cycle 11/Day 1 (n=15,24,16,15) | 1.0 [0.0 to 2.1] | 0.3 [-0.6 to 1.3] | 0.8 [0.0 to 1.6] | -0.2 [-1.6 to 1.2]
  Change at Cycle 13/Day 1 (n=13,19,15,10) | 1.1 [-0.4 to 2.7] | 0.7 [-0.2 to 1.5] | 1.3 [0.4 to 2.2] | 0.7 [-0.7 to 2.1]
  Change at Cycle 15/Day 1 (n=7,17,12,8) | 2.3 [0.8 to 3.8] | 0.9 [-0.3 to 2.0] | -0.1 [-1.4 to 1.3] | 1.3 [0.0 to 2.5]
  Change at Cycle 17/Day 1 (n=6,11,11,7) | 2.4 [0.9 to 3.8] | 0.7 [-0.7 to 2.1] | 0.7 [-1.3 to 2.6] | 2.1 [-0.1 to 4.3]
  Change at Cycle 19/Day 1 (n=6,10,9,5) | 2.1 [0.6 to 3.6] | 0.8 [-0.6 to 2.3] | 0.3 [-1.6 to 2.2] | 2.4 [1.2 to 3.7]
  Change at Cycle 21/Day 1 (n=6,9,7,4) | 1.7 [-0.3 to 3.7] | 1.0 [-1.2 to 3.2] | 0.4 [-1.0 to 1.8] | 2.1 [0.8 to 3.4]
  Change at Cycle 23/Day 1 (n=5,7,6,4) | 2.2 [0.0 to 4.4] | -0.3 [-1.3 to 0.8] | 0.9 [-1.7 to 3.4] | 1.4 [0.8 to 2.0]
  Change at Cycle 25/Day 1 (n=5,7,6,3) | 1.6 [-0.9 to 4.1] | 0.5 [-2.0 to 3.0] | -0.6 [-2.7 to 1.5] | 1.4 [0.5 to 2.3]
  Change at Cycle 27/Day 1 (n=2,7,3,3) | 1.6 [-16.4 to 19.6] | 0.9 [-2.1 to 4.0] | -1.6 [-5.7 to 2.4] | 1.3 [0.9 to 1.7]
  Change at Cycle 29/Day 1 (n=2,5,2,3) | 3.2 [-26.5 to 32.8] | 0.0 [-2.3 to 2.2] | -1.3 [-15.0 to 12.5] | 1.3 [-0.4 to 3.0]
  Change at Cycle 31/Day 1 (n=1,5,2,2) | 4.5 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | -0.5 [-2.1 to 1.0] | -0.1 [-26.6 to 26.4] | 1.2 [-3.1 to 5.4]
  Change at Cycle 33/Day 1 (n=1,3,2,1) | 4.5 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | -0.2 [-4.4 to 3.9] | -0.8 [-29.3 to 27.8] | 0.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 35/Day 1 (n=0,4,1,1 ) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [-1.9 to 1.2] | -1.2 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | 3.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 37/Day 1 (n=0,4,0,1) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.4 [-2.1 to 1.2] | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 1.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 39/Day 1 (n=0,2,0,1) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [-0.3 to -0.3] | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 2.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 41/Day 1 (n=0,2,0,1) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.2 [-2.3 to 2.0] | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 1.5 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 43/Day 1 (n=0,1,0,1) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 1.8 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 45/Day 1 (n=0,0,0,1 ) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 2.5 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable.
  Change at Cycle 47/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.2 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 49/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 51/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 53/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.2 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 55/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.3 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 57/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 0.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 59/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.2 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 61/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | 0.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 63/Day 1 (n=0,0,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at Cycle 65/Day 1 (n=0,1,0,0) | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | -0.2 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle. | NA [NA to NA] — Data was not analyzed as no participants were evaluable for the particular cycle.
  Change at end of treatment (n=21,29,26,21) | 1.3 [0.5 to 2.1] | 1.0 [0.3 to 1.6] | 1.5 [0.2 to 2.8] | 1.2 [0.0 to 2.4]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib + FOLFIRI | Bevacizumab + FOLFIRI | Axitinib + FOLFOX | Bevacizumab + FOLFOX
Serious Adverse Events (participants affected / at risk) | 17/46 | 9/51 | 11/36 | 5/35
Other Adverse Events (participants affected / at risk) | 45/46 | 51/51 | 35/36 | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + FOLFIRI (N=46) | Bevacizumab + FOLFIRI (N=51) | Axitinib + FOLFOX (N=36) | Bevacizumab + FOLFOX (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Otosalpingitis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Haemorrhagic ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 0 | 1 | 0
Disease progression (General disorders) | 2 | 3 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cellulitis pharyngeal (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + FOLFIRI (N=46) | Bevacizumab + FOLFIRI (N=51) | Axitinib + FOLFOX (N=36) | Bevacizumab + FOLFOX (N=35)
Anaemia (Blood and lymphatic system disorders) | 6 | 11 | 4 | 5
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 6 | 6 | 5 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 20 | 27 | 20 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4 | 8 | 5
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Otosalpingitis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 7 | 0 | 9 | 1
Age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 1
Asthenopia (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 1 | 0 | 1
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 2
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0
Mydriasis (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 12 | 11 | 7 | 9
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 7 | 16 | 3 | 10
Defaecation urgency (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 32 | 25 | 15 | 11
Dry mouth (Gastrointestinal disorders) | 3 | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 7 | 5 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 2 | 1 | 2
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 27 | 30 | 18 | 16
Odynophagia (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Painful defaecation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Peristalsis visible (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 6 | 2 | 1 | 0
Proctitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 3 | 0 | 3
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 11 | 7 | 9 | 7
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tooth erosion (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 22 | 18 | 12 | 3
Asthenia (General disorders) | 13 | 11 | 6 | 6
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 3 | 1 | 1
Chills (General disorders) | 2 | 1 | 2 | 2
Device occlusion (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 21 | 18 | 12 | 9
Implant site haematoma (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 7 | 11 | 4 | 3
Oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 7 | 2 | 0 | 1
Pain (General disorders) | 0 | 1 | 3 | 1
Performance status decreased (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 7 | 5 | 3
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0
Thrombosis in device (General disorders) | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 1 | 1 | 2
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 5 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Colostomy infection (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 2 | 1 | 0
Device related infection (Infections and infestations) | 1 | 1 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 1 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 5 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 3 | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 1
Anal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase (Investigations) | 1 | 0 | 0 | 3
Alanine aminotransferase increased (Investigations) | 3 | 2 | 1 | 2
Aspartate aminotransferase (Investigations) | 1 | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 1 | 2
Blood albumin decreased (Investigations) | 2 | 1 | 0 | 0
Blood alkaline phosphatase (Investigations) | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 4 | 0 | 0 | 2
Blood bilirubin (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine (Investigations) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 4 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 1 | 2
Carcinoembryonic antigen increased (Investigations) | 1 | 0 | 0 | 0
Clostridium test positive (Investigations) | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
General physical condition normal (Investigations) | 0 | 0 | 0 | 1
Haemoglobin (Investigations) | 0 | 0 | 1 | 2
Haemoglobin decreased (Investigations) | 3 | 5 | 3 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count (Investigations) | 1 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 4 | 3 | 3 | 2
Platelet count (Investigations) | 0 | 0 | 1 | 2
Platelet count decreased (Investigations) | 2 | 2 | 4 | 3
Visual field tests (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 13 | 4 | 5 | 2
Weight increased (Investigations) | 0 | 1 | 1 | 0
White blood cell count (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 2 | 0 | 1 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 24 | 16 | 13 | 7
Dehydration (Metabolism and nutrition disorders) | 7 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3 | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1
Cholinergic syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 3 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 5 | 1 | 3 | 4
Headache (Nervous system disorders) | 6 | 4 | 7 | 3
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 4 | 7 | 16
Paraesthesia (Nervous system disorders) | 0 | 2 | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 4 | 4 | 5
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Toxic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 3 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 5 | 3 | 2 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 2 | 3
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 3 | 4
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 8 | 5 | 2 | 3
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 3 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 4 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 15 | 4 | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 12 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Facial wasting (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 3 | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 3 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 17 | 8 | 24 | 6
Hypotension (Vascular disorders) | 3 | 1 | 2 | 2
Pallor (Vascular disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 2 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.